CLINICAL TRIAL: NCT06464939
Title: A Randomized, Double-blinded, Placebo-controlled, Phase 2 Study to Assess the Efficacy and Safety of Three Topical Applications of KH001 in Providing Long-term Relief From Dentin Hypersensitivity
Brief Title: Phase 2 Study of KH001 in Long-term Relief From Dentin Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HysensBio Co., Ltd (Industry)
Collaborators: The Forsyth Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KH-001-G201
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin Sensitivity; Denin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): KH001 and placebo
  Interventions: Drug: KH001; Drug: Placebo
- Group B (Experimental): KH001 and placebo
  Interventions: Drug: KH001; Drug: Placebo
- Group C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KH001 — Applications of KH001 over a 1 or 2-week period, and application of placebo
  Arms: Group A; Group B
Drug: Placebo — Applications of water for injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KH001 in subjects with dentin hypersensitivity.

DETAILED DESCRIPTION:
The study will consist of a screening period, a treatment period, and a follow-up period. The total duration of the study for each subject will be approximately 8 to 12 weeks. All subjects will be randomly assigned in a 1:1:1 ratio, with Group A, Group B and Group C.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old by the time of the screening visit
* Is in good general health as determined by the investigator
* Has at least 2 non-adjacent teeth and is diagnosed with hypersensitive

Exclusion Criteria:

* Is allergic to the active drug substance or other excipients used in the investigational product
* Has any history of alcohol or drug abuse
* Has received any treatment related to dentin hypersensitivity within 8 weeks prior to the screening visit
* Is jedged by the investigator as ineligible for participation for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Schiff sensitivity score | Baseline and Week 5
  Schiff sensitivity score 0-3 by an evaporative air

SECONDARY OUTCOMES:
Change from baseline in a Schiff sensitivity score | Baseline, Up to 8 Weeks
  Schiff sensitivity score 0-3 by an evaporative air
Change from baseline in a Tactile threshold | Baseline, Up to 8 Weeks
  Tactile threshold by yeaple probe
Change from baseline in Visual Analogue Scale | Baseline, Up to 8 Weeks
  Visual Analogue Scale by an evaporative air

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Hasturk, Principal Investigator — ADA Forsyth
Locations (2):
- United States (2):
  - ADA Forsyth, Cambridge, Massachusetts
  - Forsyth Institute, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No